CLINICAL TRIAL: NCT06012955
Title: Study on the Effect of Target-controlled Infusion of Propofol and Remifentanil for Patients Undergoing Cardiac Surgery
Brief Title: Study on the Effect of Target-controlled Infusion for General Anesthesia in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: TCI202112
Record Dates: First submitted 2023-08-20; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Mechanical Ventilation Time
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCI group: patients receiving general anesthesia using target-controlled infusion delivery system
  Interventions: Device: Target-controlled infusion (TCI) systems
- MCI group: patients receiving general anesthesia using conventional manual controlled infusion delivery

INTERVENTIONS:
Device: Target-controlled infusion (TCI) systems — Target-controlled infusion (TCI) with propofol and remifentanil was used for anesthesia induction and maintenance
  Groups: TCI group

SUMMARY:
The purpose of the study was to evaluate whether individualized general anesthesia with target-controlled infusion could help patients wake up early for extubation and reduce the incidence of postoperative complications, and to investigate the effectiveness and safety of its application in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older who underwent cardiac surgery

Exclusion Criteria:

* Mechanical ventilation support before surgery;
* Combined with any type of non-cardiac surgeries;
* Second exploratory thoracotomy after surgery;
* Died or discharged within 48 h after surgery;
* Missing clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or olderundergoing cardiac surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative mechanical ventilation | 4 weeks after surgery
  Duration of mechanical ventilation was defined as the time from the end of surgery to tracheal extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China